CLINICAL TRIAL: NCT02362802
Title: Myocardial Minimal Damage After Rapid Ventricular Pacing
Acronym: MyDate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Principal Investigator, Adnan Kastrati, MD, PD Dr. med. C. Kolb, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-015
Record Dates: First submitted 2015-02-01; First posted 2015-02-13 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Antitachycardia Pacing
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antitachycardia Pacing (Active Comparator): Implantable cardioverter defibrillator placement with Antitachycardia Pacing. Apart from that usual standard of care.
  Interventions: Device: Implantable Cardioverter Defibrillator
- No Antitachycardia Pacing (No Intervention): Implantable cardioverter defibrillator placement without Antitachycardia Pacing.
  Apart from that usual standard of care.

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator
  Arms: Antitachycardia Pacing

SUMMARY:
This study aims to investigate the impact of antitachycardia pacing ( ATP) on the myocardial tissue with respect to its potential micro damage measured by several myocardial markers, especially by high-sensitive TroponinT.

ELIGIBILITY:
Inclusion Criteria:

* All patients for de-novo implantation of a transvenous ICD (single chamber, dual chamber or cardiac resynchronization tehrapy) with left pectoral device position and planned apical location of the right ventricular defibrillation electrode.

Exclusion Criteria:

* Resuscitation, cardiac surgical procedure, acute coronary syndrome, acute myocardial infarction, coronary revascularisation, cardioversion or ablation during the past 4 weeks, if baseline high-sensitive Troponin T is elevated
* Known stenosis of coronary vessels with indication for coronary intervention or operative revascularisation
* Intracardiac thrombus or general contraindication against ventricular burst stimulation or intraoperative ICD-testing
* Atypical lead implantation with indication for defibrillation threshold testing by induction of ventricular fibrillation
* Right sided implantation of ICD
* Planned electrical cardioversion
* Lead explantation or -extraction during procedure
* Redo procedure (except of additional implantation of a right ventricular ICD lead)
* Present temporary pacemaker electrode
* ASA >= IV or NYHA IV
* Cardiogenic shock
* Pulmonary embolism, cerebrovascular insult or dialysis in the past 4 weeks
* Lack of consent of patient
* Minority of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
High sensitive Troponin | 14-20 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Result] Semmler V, Deutschmann C, Haller B, Lennerz C, Brkic A, Grebmer C, Blazek P, Weigand S, Karch M, Busch S, Kolb C. Myocardial Minimal Damage After Rapid Ventricular Pacing - the prospective randomized multicentre MyDate-Trial. Sci Rep. 2020 Mar 16;10(1):4753. doi: 10.1038/s41598-020-61625-8. PMID 32179792